CLINICAL TRIAL: NCT04816773
Title: Post Market Clinical Follow-Up Study for EVOLUTION® NitrX™ Keeled Tibia and EVOLUTION® NitrX™ CS/CR Femur With Cruciate Sacrificing Insert
Status: Enrolling by invitation | Type: Observational
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 20K001
Record Dates: First submitted 2021-03-17; First posted 2021-03-25 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Joint Diseases; Osteoarthritis; Arthritis Knee; Avascular Necrosis
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Newly or previously implanted patients: Multicenter, non-interventional prospective follow-up of newly or previously implanted subjects. Previously implanted subjects must be enrolled within 14 months of the study index surgery. Single study group with either newly or previously implanted patients with all EVOLUTION® NitrX™ components: Non-Porous Keeled Tibia, CS/CR Non-Porous Femur component, and EVOLUTION® MP CS tibial insert
  Interventions: Device: EVOLUTION® NitrX™

INTERVENTIONS:
Device: EVOLUTION® NitrX™ — EVOLUTION® NitrX™ Keeled Tibia and EVOLUTION® NitrX™ CS/CR Femur With Cruciate Sacrificing Insert

SUMMARY:
MicroPort Orthopedics Inc. (MPO) plans to market the EVOLUTION® NitrX™ Non-Porous Keeled Tibia and EVOLUTION® NitrX™ CS/CR Non-Porous Femur with the EVOLUTION® Cruciate Sacrificing (CS) Tibial Insert globally, including in the European Union (EU). MPO is conducting this post market clinical follow-up (PMCF) study to evaluate the safety and effectiveness of the EVOLUTION® NitrX™ Non-Porous Keeled Tibia and EVOLUTION® NitrX™ CS/CR Non-Porous Femur. These components are used along with the EVOLUTION® Cruciate Sacrificing (CS) Tibial Insert components that is marketed in the European Union (EU). This type of data collection is required by regulatory authorities for all TKA devices that do not have medium to long-term clinical evidence available.

ELIGIBILITY:
Inclusion Criteria:

1. Has previously undergone or currently has determined to undergo a primary TKA with the specified combination of components: EVOLUTION® NitrX™ CS/CR Non-Porous Femur, EVOLUTION® NitrX™ Non-Porous Keeled Tibia and EVOLUTION® CS Tibial Insert
2. Has previously undergone or currently has determined to undergo a primary TKA for any of the following:

   * non-inflammatory degenerative joint disease including osteoarthritis, traumatic arthritis, or avascular necrosis;
   * inflammatory degenerative joint disease including rheumatoid arthritis;
   * correction of functional deformity;
3. Willing to voluntarily sign the informed consent form
4. Willing and able to comply with the protocol, able to read and complete the required forms, and willing and able to adhere to the requirements of the protocol through the 10-year postoperative follow-up visit.
5. Previously implanted subjects must be enrolled within 14 months of their primary TKA implantation.

Prospective enrollment of a previously unimplanted contralateral knee is permitted in this study provided:

1. the specified combination of components (EVOLUTION® NitrX™ CS/CR Non-Porous Femur, EVOLUTION® NitrX™ Non-Porous Keeled Tibia and EVOLUTION® CS Tibial Insert) are used,
2. all other aspects of the Inclusion/Exclusion Criteria are satisfied,
3. enrollment does not exceed the subject count specified in the Clinical Trial Agreement, and
4. the subject agrees to a second Informed Consent document and data collection specific to the second TKA.

Bilateral subjects can have both TKAs enrolled in the study provided:

1. the specified combination of components (EVOLUTION® NitrX™ CS/CR Non-Porous Femur, EVOLUTION® NitrX™ Non-Porous Keeled Tibia and EVOLUTION® CS Tibial Insert) were implanted in both,
2. all other aspects of the Inclusion/Exclusion Criteria are satisfied,
3. enrollment does not exceed the subject count specified in the Clinical Trial Agreement, and
4. the subject agrees to a second Informed Consent document and data collection specific to the second TKA.

Bilateral implantation can occur at different time periods for the same subject.

Exclusion Criteria:

1. Skeletally immature (less than 21 years of age) at time of implantation
2. Has or had an overt infection at the time of implantation
3. Has or had a distant foci of infections (which may cause hematogenous spread to the implant site) at the time of implantation
4. Has or had a rapid disease progression as manifested by joint destruction or bone absorption apparent on roentgenogram at the time of implantation
5. Has or had inadequate neuromuscular status (e.g., prior paralysis, fusion, and/or inadequate abductor strength), poor bone stock, poor skin coverage around the joint which would make the procedure unjustifiable
6. Currently enrolled in another clinical investigation which could affect the endpoints of this protocol
7. Has documented substance abuse issues
8. Has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study
9. Currently incarcerated or has impending incarceration
10. Has a medical condition, as judged by the Investigator, that would interfere with the subject's ability to comply with the requirements of the protocol

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Single study group with either newly or previously implanted patients with all EVOLUTION® NitrX™ components: Non-Porous Keeled Tibia, CS/CR Non-Porous Femur component, and EVOLUTION® MP CS tibial insert
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2034-08 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
Component Survivorship of the EVOLUTION® NitrX™ Non-Porous Keeled Tibia | 10 years post-operative
  The primary endpoint is to evaluate component survivorship of the EVOLUTION® NitrX™ Non-Porous Keeled Tibia out to 10 years follow-up. Percentage of knees survived with no revisions or replacement at 10-year
Component Survivorship of the EVOLUTION® NitrX™ CS/CR Non-Porous Femur | 10 years post-operative
  The primary endpoint is to evaluate component survivorship of the EVOLUTION® NitrX™ CS/CR Non-Porous Femur out to 10 years follow-up. Percentage of knees survived with no revisions or replacement at 10-year.
Component Survivorship of the EVOLUTION® NitrX™ MP CS tibial inserts | 10 years post-operative
  The primary endpoint is to evaluate component survivorship of the EVOLUTION® NitrX™ MP CS tibial inserts out to 10 years follow-up. Percentage of knees survived with no revisions or replacement at 10-year.

SECONDARY OUTCOMES:
Functional Scores | 10 years post-operative
  To assess functional scores utilizing Knee Injury and Osteoarthritis Outcome Score (KOOS).
Functional Scores | 10 years post-operative
  To assess functional scores utilizing EQ-5D-5L.
Functional Scores | 10 years post-operative
  To assess functional scores utilizing Forgotten Joint Score (FJS).
Subject Satisfaction | 10 years post-operative
  To assess subject satisfaction with their TKA procedure via the Satisfaction Survey.
Radiolucencies | 10 years post-operative
  To assess the presence of radiolucencies surrounding the implanted femoral and tibial components present in each of the 17 zones.
To assess subject safety: Adverse Events | 1, 3, 5, 7, 10 years
  To assess safety of the EVOLUTION® NitrX™ system through device-related adverse event findings and/or adverse device effects during follow-up visits.
To assess device tolerability within subject: Adverse Events | 10 years post-operative
  To assess tolerability of the EVOLUTION® NitrX™ system service-related adverse event findings and/or adverse device effects during follow-up visits.

CONTACTS AND LOCATIONS:
Locations (2):
- Sah Orthopaedic Associates, Fremont, California, United States
- MSK Doctors, The Keep Clinic, Grantham, Lincolnshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No